CLINICAL TRIAL: NCT05273788
Title: Thoracic Neuromodulation for Diabetic Gastroparesis
Acronym: TNM-DGp
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1870454; Pro00146242 (Other: Medical University of South Carolina)
Record Dates: First submitted 2022-03-02; First posted 2022-03-10 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Gastroparesis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- 1Hz Arm (Active Comparator): ThorS-MagNT treatment intervention with 2400 total stimulations at 1Hz with the magnetic coil.
  Interventions: Device: 2400 ThorS-MagNT Stimulations at 1Hz
- 10Hz Arm (Active Comparator): ThorS-MagNT treatment intervention with 2400 total stimulations at 10Hz with the magnetic coil.
  Interventions: Device: 2400 ThorS-MagNT Stimulations at 10Hz
- Sham Arm (Sham Comparator): Sham intervention with 2400 total sham stimulations with the magnetic coil.
  Interventions: Device: Sham Stimulations

INTERVENTIONS:
Device: 2400 ThorS-MagNT Stimulations at 1Hz — The inferior angles of the scapula will serve as landmarks for the T7 level. A mapping procedure is performed with subject in the seated position using a single-pulse stimulation circular 90- mm coil to determine the location and minimum intensity of stimulation left and right of the T7 spinous process required to achieve a motor evoked response (MEP) of 50 μV with 50% of trials (resting motor threshold) in the upper rectus abdominis or external oblique muscles. The intensity for ThorS-MagNT is set at 150% above motor threshold. 1 Hz ThorS-MagNT, one of 4 total trains is delivered over 5 minutes with 3-min rest intervals on both right and left sides (total 1200 pulses/side).
  Arms: 1Hz Arm
Device: 2400 ThorS-MagNT Stimulations at 10Hz — The inferior angles of the scapula will serve as landmarks for the T7 level. A mapping procedure is performed with subject in the seated position using a single-pulse stimulation circular 90- mm coil to determine the location and minimum intensity of stimulation left and right of the T7 spinous process required to achieve a motor evoked response (MEP) of 50 μV with 50% of trials (resting motor threshold) in the upper rectus abdominis or external oblique muscles. The intensity for ThorS-MagNT is set at 150% above motor threshold. 10Hz ThorS-MagNT involves delivering one train of 100 pulses per minute with 50-second rest intervals over twelve minutes on both right and left sides (total 1200 pulses/side).
  Arms: 10Hz Arm
Device: Sham Stimulations — The inferior angles of the scapula will serve as landmarks for the T7 level. A mapping procedure is performed with subject in the seated position using a single-pulse stimulation circular 90- mm coil to determine the location and minimum intensity of stimulation left and right of the T7 spinous process required to achieve a motor evoked response (MEP) of 50 μV with 50% of trials (resting motor threshold) in the upper rectus abdominis or external oblique muscles. The intensity for ThorS-MagNT is set at 150% above motor threshold. Sham stimulations, one of 4 total trains is delivered over 5 minutes with 3-min rest intervals on both right and left sides (total 1200 pulses/side).
  Arms: Sham Arm

SUMMARY:
The global incidence of diabetes is rising. Gastroparesis is a significant complication of diabetes that results in debilitating symptoms and affects quality of life. Current treatment options for diabetic gastroparesis are limited. Significant visceral afferent neuropathy is associated with diabetic gastroparesis and sympathetic overactivity is seen in nausea, both type 1 and 2 diabetes, and diabetic complications. These dysfunctions can result from neuropathy affecting the thoracic spinal nerves that carry both general visceral afferents and preganglionic sympathetic efferents in the greater splanchnic nerve, innervating the foregut. Neuromodulation of the thoracic spinal nerves should improve diabetic gastroparesis symptoms and restore quality of life by improving neuropathy and gastric sensori-motor function. The investigators has developed and refined a novel, noninvasive, neuromodulation treatment, Thoracic Spinal Nerve Magnetic Neuromodulation Therapy (ThorS-MagNT). In an uncontrolled trial of adults with diabetic gastroparesis, ThorS-MagNT the investigators demonstrated feasibility, acceptability, and improvement of DGp symptoms. Whether active neuromodulation is better than sham therapy and the optimal frequency of treatment are not known. The investigators propose to conduct a dose-ranging, sham-controlled trial (pilot NIH Stage 1b) to assess the effect of ThorS-MagNT on symptom severity and quality of life in diabetic gastroparesis (TNM-DGp Trial). The investigators will test the hypothesis that ThorS-MagNT will improve visceral afferent neuropathy, autonomic and gastric dysfunction, compared to sham. The investigators will also test whether any improvements are due to neuromodulation of (a) peripheral spino-gut axis or (b) central structures of the limbic system and autonomic network, or both. Successful completion of this pilot study will provide insights into gastroparesis disease processes and inform mechanisms of action of neuromodulation therapy in addressing disruption of the brain-gut axis. Expected outcomes include development of a novel, non-invasive, safe and efficacious therapy for diabetic gastroparesis. These efforts will inform future true efficacy testing in an NIH Stage 2 trial using multiphase optimization strategy (MOST) design.

DETAILED DESCRIPTION:
The proposed TNM-DGp trial is a pilot sham-controlled RCT to test the preliminary efficacy of ThorS-MagNT to improve DGp symptom severity and related quality of life. The investigators will also explore mechanisms of change and potential moderators of treatment outcome after ThorS-MagNT. The trial will be conducted over the 3-year pilot RO1.

Randomization: Using the magnitude of change in DGp symptom severity in the initial pilot trial, the investigators will randomize 48 patients in a 1:1:1 ratio to either receive sham, 1 Hz, or 10 Hz ThorS-MagNT over a 5-day period. The investigators will use blocked randomization with a block size ranging from 3 to 6 and known only to the biostatistician. The biostatistician will create the randomization sequence for all participants prior to any pre-treatment assessments. Treatment allocation will be made available to the interventionists only after baseline assessments, determination of eligibility, and informed consent.

Participants (N = 48): The investigators will recruit TNM-DGp trial participants at Augusta University. Approximately 2-3 DGp patients are seen per week at our center. To further facilitate recruitment, advertisements will be put into newsletters of both hospitals, local newspaper, and radio. Flyers will be placed in GI, family medicine, internal medicine, and endocrine clinics, and locoregional colleagues will be emailed. Forty-eight adult, DGp outpatients with refractory symptoms of greater than 6 months and moderate-severe disease (total American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptoms Index (ANMS GCSI) score greater than or equal to 2.0) will be recruited. Participants will be screened by phone to assess eligibility and interest in the study. Those who are eligible and interested in the study will complete informed consent.

Sample size justification: Assuming a responder rate of 30% for the sham arm, we consider a 1:1:1 balanced design for the sham, 1 Hz, and 10 Hz treatment arms, respectively. For the primary clinical outcome, the difference is assessed between sham and the combined treatment arm (1 Hz and 10 Hz), giving a 1:2 allocation. A sample size of 14 per treatment arm is required to observe a responder rate of 65% for the combined treatment arm with 80% power at 5% significance level. This sample size is sufficient to observe a 1-point improvement in the PAGI-QOL score (secondary clinical outcome) with 85% power. Accounting for a 15% dropout in the study, the investigators will need 16 subjects per treatment arm. For the proposed interim analysis at 33% and 66% recruitment, the investigators will have enough sample size (5 and 10 per treatment arm respectively) to achieve 80% power if the responder rate in the treatment arms is 90% and 77% respectively.

Clinical outcome (Aim 1) measures: The primary clinical outcome will be responder rate with responder defined as ≥30% improvement in gastroparesis symptom severity by the Week 4 ANMS total GCSI-DD compared to baseline. The total ANMS GCSI-DD score includes a 7-day average of 5 gastroparesis-specific items. A greater than 30% reduction in total symptom score is defined as a responder by the FDA User Manual for the ANMS GSCI-DD. Secondary clinical outcome will be improvement in quality of life, defined by a 1-point improvement in Patient Assessment of Gastrointestinal Symptoms-Quality of Life (PAGI-QOL). ANMS GCSI-DD will be collected monthly for one year after treatment. Duration of response will be defined as time to loss of response (<30% improvement over baseline total ANMS GCSI-DD score).

Exploratory mechanisms of change (Aim 2) assessments: The investigators will evaluate potential mechanisms of change pre- to post-treatment including change in activity levels and functional connectivity to surrounding brain regions of the insula by dipolar source localization and fMRI; sensation by quantitative sensory testing (QST) and satiety test; autonomic function testing; and and gastric emptying breath tests. Exploratory moderators of outcome measures. The investigators will characterize patients at pre-treatment by various clinical variables including: age, gender, type of diabetes (type 1 vs type 2), glycemic control (Hemoglobin A1c (HbA1c)), hip/waist circumference, Body Mass Index (BMI), Gastrointestinal-specific anxiety (Visceral Sensitivity Index; (VSI)), interoceptive awareness (Multidimensional Assessment of Interoceptive Awareness, (MAIA)), Patient-Reported Outcome Measurement Information System (PROMIS), and presence of depression or anxiety (by Hospital Anxiety and Depression Scale; (HADS)). The investigators will explore these characteristics as potential moderators of treatment outcome (associated with change in total ANMS GSCI-DD and outcome questionnaire scores).

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient DGp patients with refractory symptoms and total ANMS GCSI-DD score ≥ 2.0 (moderate-severe severity) during screening period;
2. Men or women age less than 85;
3. No known mucosal disease;
4. Speak, write, and understand English (by self-report);
5. On stable doses of any medication for 30 days prior to entering the study (exceptions are psychotropic, opioids, and/or illicit drugs) and agrees not to change medications or dosages during the study period.

Exclusion Criteria:

1. Postsurgical gastroparesis;
2. Gastrointestinal obstruction;
3. Prior gastric surgery (fundoplication, gastric resection or pyloroplasty);
4. Achalasia, Chronic Intestinal Pseudo-obstruction, Colonic Inertia with one complete spontaneous bowel movement (CSBM) less than every 2 weeks;
5. Active inflammatory bowel disease;
6. Use of opioids greater than 3 times a week and marijuana more than 5 times a week;
7. Change in neuromodulator dosage in last 3 months (tricyclic antidepressants, gabapentin, olanzapine, etc.);
8. Use of sympathomimetics;
9. Seizure history or disorder;
10. Active serious psychiatric illness that would warrant independent attention;
11. Severe, unstable cardiac disease and arrhythmias;
12. Metal implants that are not MR safe, gastric electrical stimulators (GES), deep brain stimulators (DBS), sacral nerve stimulators (SNS), or pacemakers;
13. Pregnant women or nursing mothers;
14. Enteral or parenteral feeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Responder rate | 4 weeks
  Responder is defined as ≥30% reduction n gastroparesis symptom severity score by the Week 4 total ANMS GCSI-DD score compared to baseline.

SECONDARY OUTCOMES:
Quality of life (QOL) | 4 weeks
  Improvement in QOL is defined by a 1-point reduction in Patient Assessment of Gastrointestinal Symptoms-Quality of Life (PAGIQOL).

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No